CLINICAL TRIAL: NCT03788070
Title: Prevalence of Preoperative Dehydration in Major Elective Urologic Surgery and Its Impact on Postoperative Outcome
Acronym: DEHYD
Status: Terminated | Type: Observational
Why Stopped: Due to COVID-19 study inclusion was halted on March 16, 2020 after 309 days.
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: LOLD 01-19
Record Dates: First submitted 2018-12-19; First posted 2018-12-27 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Dehydration; Postoperative Nausea and Vomiting; Postoperative Complications
MeSH Terms: conditions — Dehydration; Postoperative Nausea and Vomiting; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to measure the prevalence of preoperative dehydration in elective major abdominal urologic surgery when we apply our daily standard operation procedures. Secondary objectives are to assess the impact of preoperative dehydration on postoperative outcome. The hypothesis is that preoperative dehydration leads to more postoperative complications.

DETAILED DESCRIPTION:
The information about the impact of preoperative dehydration on postoperative outcome is conflicting. One of the reported difficulties of the studies in this field is to get adequate power for statistical significance. The incidence of preoperative dehydration in different surgical populations has been reported in about one third of patients. The prevalence in the urologic population is not known.

This is a monocentric observational study with no study intervention. The goal is to consecutively include all patients undergoing major urologic surgery during 365 days who meet the inclusion criteria to assess the prevalence of preoperative dehydration in elective major abdominal urologic surgery when the standard operation procedures of the University Hospital Bern are applied.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Major elective urologic surgery i. Prostate surgery ii. Bladder surgery iii. Kidney surgery iv. Various laparotomies / laparoscopies (e.g. retroperitoneal lymphadenectomy)
* Standard procedure planned
* Standard perioperative management planned
* Informed consent

Exclusion Criteria:

* Preoperative iv-fluids
* Pregnancy (which is a contraindication to this type of surgery per se)
* Inability to give informed consent (e.g. severe psychiatric disorder, dementia)
* Inability to complete the Quality of Recovery (QoR) questionnaire
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The project population will be all patients undergoing major urologic surgery at the Department of Urology, Inselspital Bern, meeting the inclusion criteria. The number of participants depends on the amount of surgeries of patients meeting the inclusion criteria taking place during the inclusion period of 365 days.
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Dehydration at Induction of Anesthesia | Time point 0: time (estimated between 7am and 4pm on day of surgery) at Induction of Anesthesia for Major Urologic Surgery
  Number of dehydrated patients judged by urine specific gravity, osmolality, creatinine, color.

SECONDARY OUTCOMES:
Postoperative Nausea and Vomiting (PONV) | 6 hours, 24 hours and 48 hours postoperatively
  Number of patients with postoperative nausea and/or vomiting at 6, 24 and 48 hours postoperatively.
Gastrointestinal function (flatus/defecation) postoperatively | 24 hours and 48 hours postoperatively
  Time of first flatus or defecation
Renal function postoperatively | 6 hours, 24 hours and 48 hours postoperatively
  Creatinine 6, 24 and 48 hours postoperatively.
Fluid balance | within 24 hours postoperatively
  Judged by administered and lost fluids intraoperatively and by weight balance on postoperative day (POD) 1.
Complications within hospitalization | within hospital stay, expected to be within 2 weeks postoperatively
  Number of complications according to a prospective list
Quality of recovery | 24 hours postoperatively
  Changes in Quality of Recovery using the validated 15 items quality of recovery (QoR-15) score : QoR is a patient reported outcome short questionnaire that measure the quality of recovery after surgery and anaesthesia. It incorporates 5 dimensions of health (patient support, comfort, emotions, physical independence, pain). This is a shortened validated version of the QoR 40 including 15 items. QoR-15, with a score range from 0 to 150 (0 worst possible, 150 best possible), is easy to perform. Recently a meta-analysis showed that QoR 15 fulfils requirements for outcome measurement instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas M Löffel, M.D., Principal Investigator — Inselspital University Hospital Bern
Locations (1):
- Inselspital University Hospital Bern, Bern, Switzerland